CLINICAL TRIAL: NCT02790060
Title: Peur De l'Hypoglycémie et Variabilité Glycémique Chez Les Sujets Diabétiques de Type 1
Brief Title: Fear of Hypoglycemia and Glycemic Variability
Acronym: VARDIA
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VARDIA
Record Dates: First submitted 2016-02-02; First posted 2016-06-03 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-05

CONDITIONS: Type 1 Diabetes
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * blood (whole blood + plasma + serum)
  * urines
Oversight: Data Monitoring Committee: No

SUMMARY:
Subjects with type 1 diabetes are invited to provide usual blood glucose monitoring and a blood glucose profile (Pre/ post prandial Blood Glucose + Night Blood Glucose) on 3 occasions in a 2 week time period, in addition to the filling of 5 questionnaires including fear of hypoglycemia-2 questionnaire.

DETAILED DESCRIPTION:
Subjects with type 1 diabetes are invited to provide usual blood glucose monitoring and a blood glucose profile (Pre/ post prandial Blood Glucose + Night Blood Glucose) on 3 occasions in a 2 week time period, in addition to the filling of questionnaires including fear of hypoglycemia-2 questionnaire.

Biobanking of urine/blood Collection of key medical informations by investigators

Questionnaires :

* socio-economic status
* Fear of hypoglycemia-2
* Anxiety Depression scale (HAD)
* Health survey (SF36, SF12)
* Satisfaction to treatment (DHP-18)
* Dutch Eating Behavior Questionnaire (DEBQ)
* Pittsburgh quality of sleep (PSQI)
* Blood Glucose diary

ELIGIBILITY:
Inclusion Criteria :

* type 1 diabetes
* at least 2 Blood Glucose monitoring daily
* on insulin for more than 5 years

Exclusion Criteria :

* not stable metabolic condition (infection, steroid therapy)
* below 3 months change in insulin treatment
* other clinical trial
* renal failure (eDFG below 30 ml/min/1.73 m²)
* Pregnancy and/or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Fear of hypoglycemia score | 2 weeks
  hypoglycemia questionnaire and hypoglycemia reported by patients

SECONDARY OUTCOMES:
quality of life | from 2 weeks up to 3 months
  SF12 questionnaire done once at home and sent at least 2 weeks after onsite visit
Standard Deviation (SD) of recorded Home Monitoring of Blood Glucose (HMPG) | 2 weeks
  reports of 2 weeks 4 points profil of HMPG and 3 days of 7 points profil of HMPG

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - University Hospital of Tours, Tours, France
  - Angers University Hospital, Angers
  - Brest University Hospital, Brest
  - La Roche sur Yon Hospital, La Roche-sur-Yon
  - La Rochelle Hospital, La Rochelle
  - CH Bretagne sud, Lorient
  - Chu de Nantes, Nantes
  - Poitiers University Hospital, Poitiers
  - Chu de Rennes, Rennes

REFERENCES:
- [Derived] Saulnier PJ, Briet C, Gand E, Chaillous L, Dubois S, Bonnet F, Leguerrier AM, Fradet G, Delcourt Crespin I, Kerlan V, Gouet D, Perlemoine C, Ducluzeau PH, Pichelin M, Wargny M, Gonder-Frederick L, Ragot S, Hadjadj S, Cariou B; VARDIA study group. No association between fear of hypoglycemia and blood glucose variability in type 1 diabetes: The cross-sectional VARDIA study. J Diabetes Complications. 2019 Aug;33(8):554-560. doi: 10.1016/j.jdiacomp.2019.05.003. Epub 2019 May 10. PMID 31182337